CLINICAL TRIAL: NCT06457087
Title: Confocal Laser Endomicroscopy in the Diagnosis of Peripheral Pulmonary Lesions
Brief Title: Optical Biopsy for Peripheral Pulmonary Lesions
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Other Study IDs: SHCHE202402
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Peripheral Pulmonary Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with peripheral pulmonary lesions: A total of 150 patients with peripheral pulmonary lesions who meet the inclusion and exclusion criteria will be prospectively enrolled, of which 100 patients will be used for the development of CLE interpretation criteria, and 50 patients will be used for the validation of the criteria.

SUMMARY:
The purpose of the study is to describe confocal laser endomicroscopy (CLE) interpretation criteria for different types of peripheral pulmonary lesions (PPLs), with histopathological correlation, and to perform the validation of these criteria.

DETAILED DESCRIPTION:
CLE is a modern imaging technique that uses an excitation laser light to create real-time microscopic images of tissues. During transbronchial lung biopsy, CLE has the potential to provide real-time non-invasive diagnosis of PPLs ("optical biopsy"). In this study, we will obtain CLE images within the target lesion before taking a biopsy during transbronchial lung biopsy of PPLs. We will compare the results of the "optical biopsy" with the corresponding histopathological results and develop CLE interpretation criteria for different types of PPLs. In addition, we will perform the validation of these criteria to evaluate the ability of CLE to discriminate between benign and malignant PPLs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years.
2. Chest CT shows peripheral pulmonary lesions (peripheral pulmonary lesions are lesions beyond the segmental bronchi that are invisible during bronchoscopy), and transbronchial biopsy is considered necessary and feasible.
3. Patients who have good compliance and sign informed consent.

Exclusion Criteria:

1. Patients with known allergy for fluorescein.
2. Pregnant or lactating women.
3. Patients with contraindications of bronchoscopy.
4. The investigators believe that patient has other conditions that are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral pulmonary lesions scheduled for transbronchial lung biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of CLE in differential diagnosis of benign and malignant PPLs | 6 months post-procedure
  Diagnostic accuracy is defined as the number of lesions correctly identified as malignant or benign using our proposed CLE interpretation criteria divided by the total number of lesions.

SECONDARY OUTCOMES:
Sensitivity, specificity of CLE in differential diagnosis of benign and malignant PPLs | 6 months post-procedure
  Sensitivity is defined as the number of lesions correctly identified as malignant using our proposed CLE interpretation criteria divided by the total number of malignant lesions. Specificity is defined as the number of lesions correctly identified as benign using our proposed CLE interpretation criteria divided by the total number of benign lesions.
positive predictive value, and negative predictive value of CLE in differential diagnosis of benign and malignant PPLs | 6 months post-procedure
  The positive predictive value is the percentage of true malignant lesions among all lesions identified as malignant using our proposed CLE interpretation criteria. The negative predictive value is the percentage of true benign lesions among all lesions identified as benign using our proposed CLE interpretation criteria.
Diagnostic accuracy of CLE in differential diagnosis of different types of PPLs | 6 months post-procedure
  Different types of PPLs include different types of common malignant PPLs (e.g., adenocarcinoma, squamous cell carcinoma, small cell lung carcinoma, etc.) and different types of common benign PPLs (e.g., inflammation, tuberculosis, fungal infection, etc.). Diagnostic accuracy is defined as the number of lesions correctly identified as a specific disease using our proposed CLE interpretation criteria divided by the total number of lesions.
Incidence of complications | 1 month post-procedure
  Complications mean a composite of procedure related adverse advents during and after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No